CLINICAL TRIAL: NCT05861336
Title: Phase II Study of Gemcitabine Plus Nab-Paclitaxel in Combination With Losartan Followed by Stereotactic Radiotherapy for Locally Advanced Pancreatic Cancer: OVERPASS Trial
Brief Title: GEM+Nab-Paclitaxel Plus Losartan Followed by Stereotactic Radiotherapy for Locally Advanced Pancreatic Cancer
Acronym: OVERPASS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST157.04
Record Dates: First submitted 2023-03-21; First posted 2023-05-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Losartan; Gemcitabine; Taxes; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy+Losartan+Stereotactic Radiation (Experimental): Chemotherapy will be administered for six cycles as per clinical practice (nab-paclitaxel and gemcitabine: nab-paclitaxel 125 mg/m2 on days 1, 8, and 15, Gemcitabine 1000 mg/m2 on days 1, 8 and 15 every 28 days) Losartan will be administered per os every day during induction chemotherapy and maintained until starting SBRT.
  SBRT will be administered in 7 consecutive fractions for a total dose of 35-42 Gy if no progression will be observed after induction therapy.
  Interventions: Drug: Losartan; Drug: Gemcitabine; Drug: Nab paclitaxel; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Losartan — Losartan will be administered at the dose of 25 mg PO qd starting on Cycle 1 Day 1. If this dose will be tolerated during week 1, escalation to 50 mg PO qd at Cycle 1 Day 8
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 on days 1, 8 and 15 every 28 days
Drug: Nab paclitaxel — nab-paclitaxel 125 mg/m2 on days 1, 8, and 15
Radiation: Stereotactic Body Radiation Therapy — 7 consecutive fractions for a total dose of 35-42 Gy

SUMMARY:
Single-arm, prospective, phase II study to evaluate safety and activity of an induction therapy with Gemcitabine (GEM) and nab-paclitaxel plus Losartan followed by Stereotactic Radiotherapy (SBRT) in patients affected by Locally Advanced Pancreatic Cancer (LAPC).

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is a malignant disease presenting high mortality rates, with a 5-year survival of about 11%, partly because of its known resistance to Chemotherapy (CHT) and Radiotherapy (RT). Radiation therapy in locally advanced and borderline resectable pancreatic cancer improves only local control as demonstrated by 5 studies published from 1980 to 2011 and confirmed by the more recent LAP-07 trial, which investigated conventional RT after induction CHT with the same results.

Losartan was administered because it indirectly affects tumor microenvironment mechanisms of chemo- and radioresistance. PC cells, through transforming growth factor-β (TGF-β), platelet-derived growth factor (PDGF) and Angiotensin II activating signaling pathways lead to tumor microenvironment (TME) cells activation, like pancreatic stellate cells, which play a key role in chemoresistance. Angiotensin system and TGF-β increase and maintain the extracellular matrix, which acts as a barrier against drugs. Murphy et al. showed that Losartan administration during chemotherapy resulted in an effective decrease in plasma levels of TGF-β. Their unexpected successful results suggest that targeting not only tumor but also TME might be a novel treatment paradigm.

The purpose of this study is to prospectively evaluate the safety and activity, in terms of resectability rate, of GEM-nab-paclitaxel chemotherapy with concurrent Losartan followed by SBRT in patients with LAPC.

Secondary endpoints are margin-negative resection rate (R0), progression-free survival (PFS), overall survival (OS), blood biomarkers response, safety and quality of life. A Carbohydrate antigen-19.9 (CA19.9) reduction ≥15% from baseline to the end of induction therapy and Carcinoma embryonic antigen (CEA) are tested as a reliable prognostic factor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed pancreatic carcinoma
2. Clinical stage I-III, according to tumor, nodes and metastases (TNM) 8th ed.
3. Locally advanced disease, as defined per National Comprehensive Cancer Network (NCCN) Guidelines version 1.2022 (Appendix D)
4. Baseline systolic blood pressure (SBP) ≥ 100 mmHg (baseline SBP will be documented during the enrolment visit in a resting, seated position at least five minutes apart; SBP will be established as the average of the two readings; if SBP is borderline it may be measured in the other arm);
5. Age >18 years and ≤75 years.
6. Life expectancy greater than 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
8. Presence of at least one measurable lesion in agreement to RECIST 1.1 criteria
9. Patients must have normal organ and marrow function as defined below:
10. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence, prior to study entry and continuing throughout the study period and for 6 months after final study drug administration. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Clinical stage IV, according to TNM 8th ed.
2. Patients who have previously received chemotherapy or radiotherapy for pancreatic cancer.
3. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to any agent used in the study.
5. Serious concomitant systemic disorders incompatible with the study (at discretion of the investigator);
6. Patient already treated on other Losartan dosages than those prescribed by protocol or treated on other Angiotensin II Receptor Blockers (ARB) therapy for hypertension or renal protection (with diabetes) at the time of enrolment;
7. Baseline hypotension, defined as systolic BP lower than 100 mmHg on two readings obtained on two separated days prior to study enrolment.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Number of participants discontinuing study treatment due to treatment related grade≥3 non-hematological adverse event [Toxicity] | 40 months
  Toxicity-related discontinuation is defined as:
  for chemotherapy + losartan phase, discontinuation due to a treatment-related ≥grade3 non-hematological adverse event; Toxicity assessments will be done using the NCI Common Terminology Criteria for Adverse Events v 5.0.
Number of participants discontinuing study treatment due to treatment related grade≥3 adverse event [Toxicity] | 40 months
  Toxicity-related discontinuation is defined as:
  for SBRT phase, discontinuation due to a ≥grade3 Adverse Events (Enteritis, Gastritis, Malabsorption, Nausea) occurring for three consecutive days.
  Toxicity assessments will be done using the NCI Common Terminology Criteria for Adverse Events v 5.0.
Resectability rate | 40 months
  Rate of patients undergoing surgery on total patient population. Resectability will be determined by Multidisciplinary team according

SECONDARY OUTCOMES:
margin-negative resection rate (R0) | 80 months
  Rate of negative margin resection determined by final pathology of the surgical specimen
progression-free survival (PFS) | 80 months
  Progression-free survival will be defined as the time from the start date of protocol therapy to first objective documentation of progressive disease (distant or local) or death due to any cause or last tumor evaluation
overall survival (OS) | 80 months
  Overall survival will be calculated as the time from the start date of protocol therapy to date of death due to any cause or last follow-up
biomarker blood response | 80 months
  A CA19.9 reduction ≥15% from baseline to the end of induction therapy and CEA are tested as a reliable prognostic factor
Incidence of Treatment-Emergent Adverse Events [Toxicity] | 80 months
  All patient will be evaluated for toxicity using the NCI Common Terminology Criteria for Adverse Events (CTCAE v 5.0). All patients will be evaluated for toxicity after each therapy session. Toxicity analyses will be performed on all patients who received at least one dose of study treatment.
  Frequency tables will be performed for all categorical variables. Continuous variables will be presented using the median and range.
Quality of life questionnaire (QLQ) | 80 months
  Quality of Life will be measured using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire that is a patient-reported outcome measure used to assess health-related quality of life in patients undergoing cancer therapy. The scale ranging from 1-4, where 1 is labeled 'Good quality of life,' and 4 is labeled 'Bad quality of life'.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Romeo, MD, Principal Investigator — IRCCS IRST
Locations (2):
- Italy (2):
  - U.O. Radioterapia IRCCS IRST, Meldola, Forlì
  - UO Oncologia, AUSL della Romagna, Ravenna

IPD SHARING:
Plan to Share IPD: No